CLINICAL TRIAL: NCT04632719
Title: MentalPlus® for Assessment and Rehabilitation of Cognitive Functions After Remission of Symptoms of COVID-19
Brief Title: The MentalPlus® for Assessment and Rehabilitation of Cognitive Function After Remission of the Symptoms of COVID-19
Acronym: MP-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Livia Stocco Sanches Valentin, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MentalPlus®
Record Dates: First submitted 2020-11-14; First posted 2020-11-17 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Cognitive Impairment; Covid19; Cognitive Dysfunction; Depression, Anxiety; Quality of Life
MeSH Terms: conditions — Cognitive Dysfunction; COVID-19; Depression; Anxiety Disorders | interventions — Physical Examination

STUDY DESIGN:
Intervention Model Description: The study has two groups. The Study Group will be the group that was remissive for COVID-19 and has some of the mentioned comorbidities, even if controlled by drugs or treatments. The Control Group will be the group with remissive patients without the aforementioned comorbidities. We will assess whether comorbidities can worsen the impairment of cognitive functions after the remission of the symptoms of COVID-19. The purpose of the research is to verify; whether COVID-19 alone in moderate to severe cases causes cognitive impairment or whether predisposing factors for such comorbidities would cause further impairment in cognitive functions after COVID-19 contraction and remission.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Covid-19 Study Group (Experimental): The Study Group will be the group that was remiss for COVID-19 and has some of the mentioned comorbidities as asthma, cardiovascular disease, cancer even if controlled by drugs or treatments.
  Interventions: Device: The use of the MentalPlus® digital game for assessment and rehabilitation of cognitive function after remission of the symptoms of COVID-19
- Covid-19 Control Group (Active Comparator): The Control Group will be the group with remissive patients without the aforementioned comorbidities. We will assess whether comorbidities can worsen cognitive functions' impairment after the remission of the symptoms of COVID-19.
  Interventions: Device: The use of the MentalPlus® digital game for assessment and rehabilitation of cognitive function after remission of the symptoms of COVID-19

INTERVENTIONS:
Device: The use of the MentalPlus® digital game for assessment and rehabilitation of cognitive function after remission of the symptoms of COVID-19 — Cognitive assessment and rehabilitation will be carried out on volunteers who have healed from COVID-19.

SUMMARY:
This study evaluates and rehabilitates the cognitive functions of attention, memory, visual perception, language, and executive by the mentalPlus® digital game of COVID-19 surviving patients after remission of symptoms.

DETAILED DESCRIPTION:
Subjects who contracted COVID-19 and present remission of symptoms will be studied, with different age groups, illiterate or literate, of both genders and with different socio-demographic characteristics. The volunteers will be submitted to the application of MentalPlus® to assess cognitive functions and SF-8® to assess Quality of Life.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by COVID-19 with or without comorbidity for cardiovascular diseases, diabetes mellitus, hypertension, cancer, asthma between the ages of 8 and 88 years of both sexes and illiterate or literate.

Exclusion Criteria:

* Disability for the instrument's use: limitation for the mobility of the upper limbs, presence of significant mental retardation that compromises the understanding of the instructions for the use of MentalPlus®, significant lowering of visual acuity.

Ages: 8 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-11-08 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Assessment of cognitive functions after COVID-19 | 1 year
  The evaluation of cognitive functions by the digital game MentalPlus® (a scale of assessment and cognitive rehabilitation) will take place as follows: Scores range from 0 [Not improved] to 10 [fully improved] at cognitive functions memory, attention and executive after training with Scale. This game is already validated and standardized for the global population. The test takes 25 minutes to play, is playful and self-explanatory. It has twelve themes with cognitive functions: short and long-term memory; selective, alternate and concentrated attention, inhibitory control of executive function and visual perception. MentalPlus® is completely randomized in its phases and themes. Therefore, the game can be used for cognitive assessment with a single theme (25 minutes of execution) or rehabilitation on 10 more themes and a final theme for reassessment of cognitive functions.

SECONDARY OUTCOMES:
Rehabilitation of cognitive functions after COVID-19 | 1 year
  Rehabilitation of cognitive functions: executive, attention, memory, visual perception, language, after the remission of the symptoms of COVID-19. MentalPlus® will be used in order to rehabilitate the cognitive functions of patients who have dysfunctions after COVID-19. The patient will play on alternate days (every other day) a theme of the game and will be rehabilitated through its 10 themes. At the end of these 10 themes, the patient will be reassessed by the last theme of the game, comprising a total of 12 themes. Each theme lasts for 25 minutes each.

CONTACTS AND LOCATIONS:
Overall Officials: Livia S. Valentin, Ph.D, Principal Investigator — University of Sao Paulo School of Medicine; Luiz Antonio M Cesar, Ph.D, Principal Investigator — University of Sao Paulo School of Medicine; Luiz Aparecido Bortolotto, Ph.D, Principal Investigator — University of Sao Paulo School of Medicine
Locations (2):
- Brazil (2):
  - Livia Stocco Sanches Valentin, São Paulo, São Paulo
  - Livia Stocco Sanches Valentin, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
The study will be shared with researchers from international centers. Therefore, the information will be made available between centers so that everyone can follow the same research protocol.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months
Access Criteria: Access will be made available by MentalPlus® APP and email.

REFERENCES:
- [Background] Beigel JH, Tomashek KM, Dodd LE, Mehta AK, Zingman BS, Kalil AC, Hohmann E, Chu HY, Luetkemeyer A, Kline S, Lopez de Castilla D, Finberg RW, Dierberg K, Tapson V, Hsieh L, Patterson TF, Paredes R, Sweeney DA, Short WR, Touloumi G, Lye DC, Ohmagari N, Oh MD, Ruiz-Palacios GM, Benfield T, Fatkenheuer G, Kortepeter MG, Atmar RL, Creech CB, Lundgren J, Babiker AG, Pett S, Neaton JD, Burgess TH, Bonnett T, Green M, Makowski M, Osinusi A, Nayak S, Lane HC; ACTT-1 Study Group Members. Remdesivir for the Treatment of Covid-19 - Final Report. N Engl J Med. 2020 Nov 5;383(19):1813-1826. doi: 10.1056/NEJMoa2007764. Epub 2020 Oct 8. PMID 32445440
- [Background] Beigel JH, Tomashek KM, Dodd LE. Remdesivir for the Treatment of Covid-19 - Preliminary Report. Reply. N Engl J Med. 2020 Sep 3;383(10):994. doi: 10.1056/NEJMc2022236. Epub 2020 Jul 10. No abstract available. PMID 32649078
- [Background] Collins FS, Stoffels P. Accelerating COVID-19 Therapeutic Interventions and Vaccines (ACTIV): An Unprecedented Partnership for Unprecedented Times. JAMA. 2020 Jun 23;323(24):2455-2457. doi: 10.1001/jama.2020.8920. No abstract available. PMID 32421150
- [Background] Benussi A, Pilotto A, Premi E, Libri I, Giunta M, Agosti C, Alberici A, Baldelli E, Benini M, Bonacina S, Brambilla L, Caratozzolo S, Cortinovis M, Costa A, Cotti Piccinelli S, Cottini E, Cristillo V, Delrio I, Filosto M, Gamba M, Gazzina S, Gilberti N, Gipponi S, Imarisio A, Invernizzi P, Leggio U, Leonardi M, Liberini P, Locatelli M, Masciocchi S, Poli L, Rao R, Risi B, Rozzini L, Scalvini A, Schiano di Cola F, Spezi R, Vergani V, Volonghi I, Zoppi N, Borroni B, Magoni M, Pezzini A, Padovani A. Clinical characteristics and outcomes of inpatients with neurologic disease and COVID-19 in Brescia, Lombardy, Italy. Neurology. 2020 Aug 18;95(7):e910-e920. doi: 10.1212/WNL.0000000000009848. Epub 2020 May 22. PMID 32444493
- [Background] Pilotto A, Benussi A, Libri I, Masciocchi S, Poli L, Premi E, Alberici A, Baldelli E, Bonacina S, Brambilla L, Benini M, Caratozzolo S, Cortinovis M, Costa A, Cotti Piccinelli S, Cottini E, Cristillo V, Delrio I, Filosto M, Gamba M, Gazzina S, Gilberti N, Gipponi S, Giunta M, Imarisio A, Liberini P, Locatelli M, Schiano F, Rao R, Risi B, Rozzini L, Scalvini A, Vergani V, Volonghi I, Zoppi N, Borroni B, Magoni M, Leonardi M, Zanusso G, Ferrari S, Mariotto S, Pezzini A, Gasparotti R, Paolillo C, Padovani A. COVID-19 impact on consecutive neurological patients admitted to the emergency department. J Neurol Neurosurg Psychiatry. 2021 Feb;92(2):218-220. doi: 10.1136/jnnp-2020-323929. Epub 2020 Oct 14. No abstract available. PMID 33055146
- [Background] Laurendon T, Radulesco T, Mugnier J, Gerault M, Chagnaud C, El Ahmadi AA, Varoquaux A. Bilateral transient olfactory bulb edema during COVID-19-related anosmia. Neurology. 2020 Aug 4;95(5):224-225. doi: 10.1212/WNL.0000000000009850. Epub 2020 May 22. No abstract available. PMID 32444492
- [Background] Brun G, Hak JF, Coze S, Kaphan E, Carvelli J, Girard N, Stellmann JP. COVID-19-White matter and globus pallidum lesions: Demyelination or small-vessel vasculitis? Neurol Neuroimmunol Neuroinflamm. 2020 May 22;7(4):e777. doi: 10.1212/NXI.0000000000000777. Print 2020 Jul. No abstract available. PMID 32444427
- [Background] Rabano-Suarez P, Bermejo-Guerrero L, Mendez-Guerrero A, Parra-Serrano J, Toledo-Alfocea D, Sanchez-Tejerina D, Santos-Fernandez T, Folgueira-Lopez MD, Gutierrez-Gutierrez J, Ayuso-Garcia B, Gonzalez de la Aleja J, Benito-Leon J. Generalized myoclonus in COVID-19. Neurology. 2020 Aug 11;95(6):e767-e772. doi: 10.1212/WNL.0000000000009829. Epub 2020 May 21. PMID 32439821
- [Background] Berger M, Terrando N, Smith SK, Browndyke JN, Newman MF, Mathew JP. Neurocognitive Function after Cardiac Surgery: From Phenotypes to Mechanisms. Anesthesiology. 2018 Oct;129(4):829-851. doi: 10.1097/ALN.0000000000002194. PMID 29621031
- [Background] Samieri C, Perier MC, Gaye B, Proust-Lima C, Helmer C, Dartigues JF, Berr C, Tzourio C, Empana JP. Association of Cardiovascular Health Level in Older Age With Cognitive Decline and Incident Dementia. JAMA. 2018 Aug 21;320(7):657-664. doi: 10.1001/jama.2018.11499. PMID 30140876
- [Background] Murray SG, Yazdany J, Kaiser R, Criswell LA, Trupin L, Yelin EH, Katz PP, Julian LJ. Cardiovascular disease and cognitive dysfunction in systemic lupus erythematosus. Arthritis Care Res (Hoboken). 2012 Sep;64(9):1328-33. doi: 10.1002/acr.21691. PMID 22549897
- [Background] Motter JN, Devanand DP, Doraiswamy PM, Sneed JR. Clinical Trials to Gain FDA Approval for Computerized Cognitive Training: What Is the Ideal Control Condition? Front Aging Neurosci. 2016 Nov 2;8:249. doi: 10.3389/fnagi.2016.00249. eCollection 2016. No abstract available. PMID 27853432
- [Background] Biessels GJ, Despa F. Cognitive decline and dementia in diabetes mellitus: mechanisms and clinical implications. Nat Rev Endocrinol. 2018 Oct;14(10):591-604. doi: 10.1038/s41574-018-0048-7. PMID 30022099
- [Background] Kim HG. Cognitive dysfunctions in individuals with diabetes mellitus. Yeungnam Univ J Med. 2019 Sep;36(3):183-191. doi: 10.12701/yujm.2019.00255. Epub 2019 Jul 24. PMID 31620632
- [Background] Duarte-Garcia A, Romero-Diaz J, Juarez S, Cicero-Casarrubias A, Fragoso-Loyo H, Nunez-Alvarez C, Llorente L, Sanchez-Guerrero J. Disease activity, autoantibodies, and inflammatory molecules in serum and cerebrospinal fluid of patients with Systemic Lupus Erythematosus and Cognitive Dysfunction. PLoS One. 2018 May 3;13(5):e0196487. doi: 10.1371/journal.pone.0196487. eCollection 2018. PMID 29723220
- [Background] Kalaria RN, Akinyemi R, Ihara M. Stroke injury, cognitive impairment and vascular dementia. Biochim Biophys Acta. 2016 May;1862(5):915-25. doi: 10.1016/j.bbadis.2016.01.015. Epub 2016 Jan 22. PMID 26806700
- [Background] Edelmann F, Stahrenberg R, Gelbrich G, Durstewitz K, Angermann CE, Dungen HD, Scheffold T, Zugck C, Maisch B, Regitz-Zagrosek V, Hasenfuss G, Pieske BM, Wachter R. Contribution of comorbidities to functional impairment is higher in heart failure with preserved than with reduced ejection fraction. Clin Res Cardiol. 2011 Sep;100(9):755-64. doi: 10.1007/s00392-011-0305-4. Epub 2011 Mar 17. PMID 21416189
- [Background] Castellino SM, Ullrich NJ, Whelen MJ, Lange BJ. Developing interventions for cancer-related cognitive dysfunction in childhood cancer survivors. J Natl Cancer Inst. 2014 Jul 30;106(8):dju186. doi: 10.1093/jnci/dju186. Print 2014 Aug. PMID 25080574
- [Background] Gottesman RF, Hillis AE. Predictors and assessment of cognitive dysfunction resulting from ischaemic stroke. Lancet Neurol. 2010 Sep;9(9):895-905. doi: 10.1016/S1474-4422(10)70164-2. PMID 20723846
- [Background] Lai CC, Shih TP, Ko WC, Tang HJ, Hsueh PR. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and coronavirus disease-2019 (COVID-19): The epidemic and the challenges. Int J Antimicrob Agents. 2020 Mar;55(3):105924. doi: 10.1016/j.ijantimicag.2020.105924. Epub 2020 Feb 17. PMID 32081636
- [Background] Wu P, Hao X, Lau EHY, Wong JY, Leung KSM, Wu JT, Cowling BJ, Leung GM. Real-time tentative assessment of the epidemiological characteristics of novel coronavirus infections in Wuhan, China, as at 22 January 2020. Euro Surveill. 2020 Jan;25(3):2000044. doi: 10.2807/1560-7917.ES.2020.25.3.2000044. PMID 31992388
- [Background] Sun P, Lu X, Xu C, Sun W, Pan B. Understanding of COVID-19 based on current evidence. J Med Virol. 2020 Jun;92(6):548-551. doi: 10.1002/jmv.25722. Epub 2020 Mar 5. PMID 32096567
- [Background] Cortegiani A, Ingoglia G, Ippolito M, Giarratano A, Einav S. A systematic review on the efficacy and safety of chloroquine for the treatment of COVID-19. J Crit Care. 2020 Jun;57:279-283. doi: 10.1016/j.jcrc.2020.03.005. Epub 2020 Mar 10. PMID 32173110
- [Background] Cortegiani A, Ippolito M, Ingoglia G, Iozzo P, Giarratano A, Einav S. Update I. A systematic review on the efficacy and safety of chloroquine/hydroxychloroquine for COVID-19. J Crit Care. 2020 Oct;59:176-190. doi: 10.1016/j.jcrc.2020.06.019. Epub 2020 Jul 11. PMID 32683212
- [Background] Li YC, Bai WZ, Hashikawa T. The neuroinvasive potential of SARS-CoV2 may play a role in the respiratory failure of COVID-19 patients. J Med Virol. 2020 Jun;92(6):552-555. doi: 10.1002/jmv.25728. Epub 2020 Mar 11. PMID 32104915
- [Background] Li YC, Bai WZ, Hashikawa T. Response to Commentary on "The neuroinvasive potential of SARS-CoV-2 may play a role in the respiratory failure of COVID-19 patients". J Med Virol. 2020 Jul;92(7):707-709. doi: 10.1002/jmv.25824. Epub 2020 Apr 10. PMID 32246783
- [Background] Chigr F, Merzouki M, Najimi M. Comment on "The neuroinvasive potential of SARS-CoV-2 may play a role in the respiratory failure of COVID-19 patients". J Med Virol. 2020 Jul;92(7):703-704. doi: 10.1002/jmv.25960. Epub 2020 May 22. PMID 32352575
- [Background] Asadi-Pooya AA, Simani L. Central nervous system manifestations of COVID-19: A systematic review. J Neurol Sci. 2020 Jun 15;413:116832. doi: 10.1016/j.jns.2020.116832. Epub 2020 Apr 11. PMID 32299017
- [Background] Valentin LS, Pietrobon R, Aguiar Junior Wd, Rios RP, Stahlberg MG, Menezes IV, Osternack-Pinto K, Carmona MJ. Definition and application of neuropsychological test battery to evaluate postoperative cognitive dysfunction. Einstein (Sao Paulo). 2015 Jan-Mar;13(1):20-6. doi: 10.1590/S1679-45082015AO3152. PMID 25993064
- [Background] Blumberg FC, Fisch SM. Introduction: digital games as a context for cognitive development, learning, and developmental research. New Dir Child Adolesc Dev. 2013 Spring;2013(139):1-9. doi: 10.1002/cad.20026. PMID 23483688
- [Background] Green CS, Bavelier D. Learning, attentional control, and action video games. Curr Biol. 2012 Mar 20;22(6):R197-206. doi: 10.1016/j.cub.2012.02.012. PMID 22440805
- [Background] Fernandez-Aranda F, Jimenez-Murcia S, Santamaria JJ, Gunnard K, Soto A, Kalapanidas E, Bults RG, Davarakis C, Ganchev T, Granero R, Konstantas D, Kostoulas TP, Lam T, Lucas M, Masuet-Aumatell C, Moussa MH, Nielsen J, Penelo E. Video games as a complementary therapy tool in mental disorders: PlayMancer, a European multicentre study. J Ment Health. 2012 Aug;21(4):364-74. doi: 10.3109/09638237.2012.664302. Epub 2012 May 1. PMID 22548300
- [Background] Oei AC, Patterson MD. Enhancing cognition with video games: a multiple game training study. PLoS One. 2013;8(3):e58546. doi: 10.1371/journal.pone.0058546. Epub 2013 Mar 13. PMID 23516504
- [Background] Boot WR, Blakely DP, Simons DJ. Do action video games improve perception and cognition? Front Psychol. 2011 Sep 13;2:226. doi: 10.3389/fpsyg.2011.00226. eCollection 2011. PMID 21949513
- [Background] Fissler P, Kolassa IT, Schrader C. Educational games for brain health: revealing their unexplored potential through a neurocognitive approach. Front Psychol. 2015 Jul 24;6:1056. doi: 10.3389/fpsyg.2015.01056. eCollection 2015. PMID 26257697
- [Background] 26. Valentin LSS, Valentin TSS, Carmona MJC, Aguilar G, Pires VY, Garcia RC, et al. Digital Game Test Neuropsychology. Fundação Biblioteca Nacional. 2014.
- [Background] 27. Valentin LSS, Valentin TSS, Carmona MJC, Garcia RC, Correa RD, Gondim GB, et al. Mental Plus. INPI - Instituto Nacional da Propriedade Intelectual. 2014.
- [Background] 28. KIRKWOOD, B. R. and STERNE, J. A. C (2006). Essential medical statistics. 2nd ed. Blackwell Science: Massachusetts, USA. p.502.
- [Background] 29. McCULLAGH, P. and NELDER, J. A., (1989). Generalized linear models. 2nd ed. Chapman and Hall: New York, USA. p.511.
- [Background] Pereira VFA, Valentin LSS. The MentalPlus(R) Digital Game Might Be an Accessible Open Source Tool to Evaluate Cognitive Dysfunction in Heart Failure with Preserved Ejection Fraction in Hypertensive Patients: A Pilot Exploratory Study. Int J Hypertens. 2018 Aug 6;2018:6028534. doi: 10.1155/2018/6028534. eCollection 2018. PMID 30174949